CLINICAL TRIAL: NCT04012398
Title: Cross-cultural Validation of the German Version of the Amsterdam Instrumental Activities of Daily Living Questionnaire® in Elderly People With and Without Mild Neurocognitive Disorder
Brief Title: Validation of the German Version of the Amsterdam Instrumental Activities of Daily Living Questionnaire®
Status: Completed | Type: Observational
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Marina Bruderer, Principal Investigator, Zurich University of Applied Sciences
Other Study IDs: A-IADL-G Validation
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Amsterdam IADL Questionnaire short, German version — Questionnaire to assess impairments in instrumental activities of daily living

SUMMARY:
Pretest and validation of the German version of the Amsterdam instrumental activities of daily living questionaire short in elderly people with normal cognition, mild cognitive impairment (MCI) or mild dementia in the German speaking part of Switzerland.

The aim is to investigate the psychometric properties of the final Amsterdam instrumental activities of daily living questionaire short (A-IADL-Q-SV) German.

Participants with normal cognition will be recruited in the community and participants with MCI and mild dementia in three memory clinic settings.

DETAILED DESCRIPTION:
Pretest:

Initially, five clinicians in the field will be asked to give feedback on the A-IADL-Q-SV German. Issues that need to be discussed include clarity of 1) answer options 2) the gradient of difficulty 3) activities or sentences. Adjustments will be made if necessary and documented.

At least five knowledgeable informants will then complete the A-IADL-Q-SV while thinking out loud and are asked to write down comments and issues on 1) the relevance of all items, 2) the applicability / meaning of the activities in Switzerland and 3) the understandability of the questions. The results will be reviewed in order to identify whether translation modifications will be necessary (e.g. rewording of items/response options). Additionally, the completed questionnaires will be explored to detect high proportions of missing items or single responses. If adjustments will be made, they will be discussed with the developer to finalize the translated German version.

Validation:

The A-IADL-Q-SV German will be tested in the community (people with normal cognition)and three memory clinic settings (people with MCI, mild dementia) including a total of 100 informants from people with normal cognition, MCI and mild dementia.

Construct validity will be assessed whether the A-IADL-Q-SV German shows the expected correlations with the mini mental state examination (MMSE), the cumulative dementia rating (CDR), the Lawton Brody Scale, the IQCODE and the Depression im Alter scale (DIA-S) Internal consistency will be assessed using item response theory (IRT) by investigating whether the translated version fits the graded response model of the original version and whether the assumptions of IRT are still met (unidimensionality, local independence and monotonicity).

Measurement invariance will be investigated using IRT by investigating whether differential item functioning is present in the comparison of the item characteristic curves of the original and translated version.

Responsiveness will be examined whether the A-IADL-Q-SV is able to discriminate people with MCI from people with normal cognition/ mild dementia Test-Retest reliability will be assessed on item level

ELIGIBILITY:
Inclusion Criteria:

* Living in the community
* Ability to understand the purpose of the study and to consent
* Knowledgeable informant available
* Signed informed consent to participate in the study

Exclusion Criteria:

* Moderate and severe cognitive decline (MMSE < 20) (people with MCI, mild dementia)
* Cognitive decline suspect based on telephone screening (people with normal cognition)
* Cognitive decline due to other causes than Alzheimer's disease, vascular dementia (e.g. neurological diseases, trauma, delirium)
* Diagnosed Depression
* Diagnosed Alcohol or Drug Misuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly community-dwelling people with normal cognition, mild cognitive impairment or mild dementia
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Amsterdam IADL Questionnaire short German version | Baseline
  Impairment in instrumental activities of daily living. Based on item response theory (IRT) the latent trait score is calculated with a mean of zero and standard deviation of one. The resulting score ranges from 20 to 80 with lower scores indicating poorer performance.
Change from baseline on the Amsterdam IADL Questionnaire short German version at two to four weeks | Follow-up after two to four weeks
  Impairment in instrumental activities of daily living. Based on item response theory (IRT) the latent trait score is calculated with a mean of zero and standard deviation of one. The resulting score ranges from 20 to 80 with lower scores indicating poorer performance.

SECONDARY OUTCOMES:
Mini Mental State Examination | Baseline
  Assessment of global cognition. The summary score ranges from 0 to 30 with higher scores indicating better performance.
Cumulative Dementia Rating | Baseline
  Assessment to stage the severity of dementia. The scoring ranges from 0 to 3 (0 = normal; 0.5 = very mild dementia; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia). Based on an interview (patient and / or relative) six domains of cognitive and functional performance (memory, orientation, judgment / problem solving, community affairs, home / hobbies and personal care.) are rated on a 5-point scale, based on this information the dementia rating is computed.
Lawton Brody Instrumental Activities of Daily Living Scale | Baseline
  The summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias
Informant Questionnaire for Cognitive Decline in the Elderly (IQCODE) short | Baseline
  Assessment to detect cognitive decline. Scores on each question (score 1 = "much better" to 5 = "much worse") are added up and devided by the number of questions. The score ranges from 1 to 5, a score of 3 means "no change", a score of 4 means "a little worse" and a score of 5 means "much worse".
Depression im Alter Scale (DIA-S) | Baseline
  The summary score ranges from 0 to 10. 0 to 2 points inconspicuous mood; > 3 points suspicious depression; > 4 points probable pathological depression

CONTACTS AND LOCATIONS:
Overall Officials: Karin Niedermann, PhD, Principal Investigator — Zurich University of Applied Sciences Zurich
Locations (1):
- Memory Clinic, Geriatrische Klinik St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruderer-Hofstetter M, Dubbelman MA, Meichtry A, Koehn F, Munzer T, Jutten RJ, Scheltens P, Sikkes SAM, Niedermann K. Cross-cultural adaptation and validation of the Amsterdam Instrumental Activities of Daily Living questionnaire short version German for Switzerland. Health Qual Life Outcomes. 2020 Oct 2;18(1):323. doi: 10.1186/s12955-020-01576-w. PMID 33008394